CLINICAL TRIAL: NCT06527365
Title: An Open-Label Multi-Dose Study to Evaluate the Safety and Efficacy of VDPHL01 in Male and Female Subjects With Androgenetic Alopecia
Brief Title: Safety and Efficacy of VDPHL01 in Males and Females With AGA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Veradermics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 250-13951-207
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Androgenetic Alopecia; AGA; Male Pattern Baldness
Keywords: Hair Loss; Male Hair Loss; Female Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Males will not be randomized. Females will be assigned once a day or twice a day treatment in an alternating fashion at each site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VDPHL01 Tablet (Experimental)
  Interventions: Drug: VDPHL01

INTERVENTIONS:
Drug: VDPHL01 — VDPHL01 Extended Release (ER) Tablet

SUMMARY:
This study will evaluate the safety and efficacy of VDPHL01 in male and female subjects with Androgenetic Alopecia (AGA).

AGA (or pattern of hair loss) is a genetic disorder caused by an excessive (too much) hair follicle response to androgens (hormone) that causes hair loss. VDPHL01 8.5 mg Tablets for males and VDPHL01 4.5 mg Tablets for females are an investigational oral drug to treat male and female pattern baldness.

This multiple center, open-label, study will last about 13 months and includes 11 study visits (screening, baseline (day 1), week 2, month 1, month 2, month 4, month 6, month 8, month 10, month 12, month 13). Male subjects that meet the study eligibility criteria will be administered VDPHL01 once daily for 12 months. Female subjects that meet the study eligibility criteria will be administered VDPHL01 either once or twice daily for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or non-pregnant female aged 18-65 years old;
* Subject has a clinical diagnosis of mild to moderate AGA;
* Subject is in good general health and has normal renal and hepatic function;
* Subject is willing to maintain at least 1/4 inch length hair during the study with the same hairstyle, hair length, and hair color throughout the study; maintain consistent use of general hair care products and regimen through the entire study;
* Subject is willing and able to administer the test article as directed read, understand, and complete required questionnaires in English;
* Subject agrees to have a micro dot tattoo placed on their scalp;
* Subject agrees to have this area photographed at study visits as indicated in the protocol.

Exclusion Criteria:

* Subject has uncontrolled blood pressure;
* Subject has symptoms or history of certain heart or thyroid conditions;
* Subject has a history of cardiac and/or thyroid diseases;
* Subject has received an organ transplant;
* Subject has a history of prescription drug abuse or illicit drug use within 6 months of screening; history of alcohol abuse within 6 months prior to screening;
* Subject has a current or recent history of dietary or weight changes;
* Subject has been diagnosed with COVID-19 within 16 weeks of baseline;
* Subject has used any topical scalp treatments for hair growth within 4 weeks prior to screening;
* Subject has had any scalp procedures, including surgical, laser, light or energy treatments, micro-needling, etc. within 6 months prior to screening;
* Subject has had previous radiation of the scalp;
* Subject has used systemic cimetidine, ketoconazole, diazoxide, or corticosteroids (including intramuscular, intraarticular, and intralesional injections) within 12 weeks prior to screening;
* Subject has used systemic beta blockers within 12 weeks prior to screening;
* Subject is currently enrolled in an investigational drug, biologic, or device study or has used an investigational treatment within 30 days prior to screening;
* Subject has used any other therapy with any medication either topical or oral that might, in the investigator's opinion, interfere with the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Changes in non-vellus Total Area Hair Count (TAHC) | Month 12
  Change from baseline in non-vellus TAHC using digital image analysis at Month 12.
Subjects Evaluation of Treatment Benefit | Month 12
  Subjects will rate their treatment benefit by responding to a hair assessment scale. The proportion of subjects by each response category will be reported at Month 12.

CONTACTS AND LOCATIONS:
Overall Officials: Reid Waldman, M.D., Study Chair — Veradermics, Inc.; Timothy Durso, M.D., Study Director — Veradermics, Inc.
Locations (4):
- United States (4):
  - 01, San Diego, California
  - 04, New Albany, Indiana
  - 03, Hackensack, New Jersey
  - 02, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: Undecided